CLINICAL TRIAL: NCT06448065
Title: A Reliability Study of Gait Classification in Children With Cerebral Palsy
Brief Title: Gait Classification in Children With Cerebral Palsy, a Reliability Study
Acronym: GCP
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K00005123
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; gait pattern classification
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adults with cerebral palsy: Children and adults with cerebral palsy who attented the gait lab for a gait analysis are included in this study.

SUMMARY:
The goal of this observational study is to assess whether gait classification patterns can be reliably obtained from video recordings in comparison with three-dimensional kinematic data.

The main questions it aims to answer are:

Are gait classifications from video recordings reliable between raters? Are gait classifications from video recordings valid in comparison with three-dimensional kinematic data?

Gait analysis data from participants who visited the gait lab in the Karolinska Hospital will be used for this purpose.

DETAILED DESCRIPTION:
Current retrospective observational study aims to assess the reliability and validity of gait pattern classification systems in ambulatory children with CP. Gait classification is often performed using kinematic gait data obtained via a three dimensional (3D) data captured in a specialized gait lab using infra-red cameras. However, not all hospitals and clinical centers have access to such a specialized gait lab, and therefore often use video recordings as an alternative for gait classification. It is currently not known whether such a classification based on solely video recordings is equally reliable in comparison with kinematic gait data. For this purpose, current study aims to assess the reliability and validity of video recordings to classify children with CP according to predefined gait classifications. Sagittal plane video recordings during barefoot walking in children with CP will be used to classify the study participants into seven different gait classification patterns. For reliability, inter-rater reliability between raters scoring the video recordings will be assessed. To evaluate whether video recordings could serve as a valid alternative for kinematic gait data, the agreement between the classifications from the video recordings and the kinematic data additionally will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis of spastic cerebral palsy
* Age 3 to 18 at the time of gait analysis
* Availability of barefoot walking data collected at the Karolinska Hospital gait lab
* Written informed consent of both parents to use the clinically collected data as research data

Exclusion Criteria:

* Main diagnosis of dyskinetic or ataxic cerebral palsy
* No barefoot walking trials available
* No kinematic data available
* BTX-A injections 6 months prior to gait analysis
* Orthopaedic surgery one year prior to gait analysis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population from which the study participants are recruited are ambulatory children and young adults with cerebral palsy. All individuals with cerebral palsy that visited the gait lab over the past 20 years are eligible to be included in the current study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability | approximately 12 months
  Assess inter-rater reliability between multiple raters assessing video recordings of gait in children with cerebral palsy
Concurrent validity | approximately 12 months
  Assess concurrent validity between outcome classifications from video recordings and from three-dimensional gait kinematics children with cerebral palsy

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Lidbeck, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No